CLINICAL TRIAL: NCT02751814
Title: Physical Activity and Screen-Time Regulations in Childcare Centers: Influence on Young Children's Health Behaviors (Pause & Play) - Aim 2
Brief Title: Physical Activity and Screen-Time Regulations in Childcare Centers - Aim 2
Acronym: Pause and Play
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Amanda Staiano, PBRC Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2015-038; U54MD008602-P02UAB (Other Grant/Funding Number: UAB); U54MD008602 (NIH)
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Results first posted 2023-12-14 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Childhood Obesity
Keywords: Childcare Center Regulations; Physical Activity; Sedentary Behavior; Screen-time Behavior
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective is to examine the physical activity and screen-time behaviors of children enrolled in licensed childcare centers before and after the enactment of new state regulations.

DETAILED DESCRIPTION:
Pause and Play aims to enroll 266 children. Each child will participate in the study for approximately 1 year. Surveys, anthropometric measures, and screen-time observations will take approximately 1 day each to complete, and the child will be given an accelerometer to wear at home for 7 days at both baseline and 1 year follow-up. Fundamental motor skill assessments will take place at baseline and 1 year follow-up after the 7 days of accelerometer wear. Staff members will spend approximately 2 weeks at each childcare center at baseline and 1 year follow-up to complete study procedures with each child.

ELIGIBILITY:
Inclusion Criteria:

* A child who is 3 or 4 years old
* Child spends at least 6 hours per day, 5 days per week at a participating childcare center
* Child will continue to attend the same childcare center for the next year

Exclusion Criteria:

* Parent/legal guardian is unwilling to provide written informed consent

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Ten licensed DOE Class A or B childcare centers will be randomly selected from a list of all DOE licensed childcare centers in East Baton Rouge Parish (EBR). From the ten centers, 266 children and their parent(s) will be recruited to complete additional measures of physical activity and screen-time behaviors.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Staiano, PhD, Principal Investigator — PBRC Assistant Professor
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Staiano AE, Allen AT, Fowler W, Gustat J, Kepper MM, Lewis L, Martin CK, Romain JS, Webster EK. State Licensing Regulations on Screen Time in Childcare Centers: An Impetus for Participatory Action Research. Prog Community Health Partnersh. 2018;12(1S):101-109. doi: 10.1353/cpr.2018.0025. PMID 29755053
- [Result] Staiano AE, Webster EK, Allen AT, Jarrell AR, Martin CK. Screen-Time Policies and Practices in Early Care and Education Centers in Relationship to Child Physical Activity. Child Obes. 2018 Aug/Sep;14(6):341-348. doi: 10.1089/chi.2018.0078. PMID 30199286
- [Result] Kracht CL, Webster EK, Staiano AE. A natural experiment of state-level physical activity and screen-time policy changes early childhood education (ECE) centers and child physical activity. BMC Public Health. 2020 Mar 24;20(1):387. doi: 10.1186/s12889-020-08533-8. PMID 32209069
- [Result] Joseph ED, Kracht CL, St Romain J, Allen AT, Barbaree C, Martin CK, Staiano AE. Young Children's Screen Time and Physical Activity: Perspectives of Parents and Early Care and Education Center Providers. Glob Pediatr Health. 2019 Jul 24;6:2333794X19865856. doi: 10.1177/2333794X19865856. eCollection 2019. PMID 31384633
- [Result] Webster EK, Martin CK, Staiano AE. Fundamental motor skills, screen-time, and physical activity in preschoolers. J Sport Health Sci. 2019 Mar;8(2):114-121. doi: 10.1016/j.jshs.2018.11.006. Epub 2018 Nov 24. PMID 30997257
- [Result] Martins, C., Webster, E. K., Bandeira, P. F. R., & Staiano, A. E. (2022). Identifying Fundamental Motor Skills Building Blocks in Preschool Children From Brazil and the United States: A Network Analysis. Journal of Motor Learning and Development, 10(1), 96-115. Retrieved Mar 27, 2024, from https://doi.org/10.1123/jmld.2021-0022
- [Result] Kracht CL, Webster EK, Staiano AE. Relationship between the 24-Hour Movement Guidelines and fundamental motor skills in preschoolers. J Sci Med Sport. 2020 Dec;23(12):1185-1190. doi: 10.1016/j.jsams.2020.06.021. Epub 2020 Jul 5. PMID 32653249
- [Result] Kracht CL, Webster EK, Staiano AE. Sociodemographic Differences in Young Children Meeting 24-Hour Movement Guidelines. J Phys Act Health. 2019 Oct 1;16(10):908-915. doi: 10.1123/jpah.2019-0018. Epub 2019 Sep 6. PMID 31491748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from 10 local preschool centers. Parents were not recruited or enrolled in this study, but they did complete surveys to assess for efficacy.
Groups:
- ECE Center Changes Between Baseline and Follow-up: Assessed differences in total EPAO score at baseline, follow-up, and overall change by policy engagement category (no engagement, some engagement, high engagement).
Period: Overall Study
Arm/Group | ECE Center Changes Between Baseline and Follow-up
Started | 175
Completed Baseline Assessments | 112
Completed | 130 (Of the 130 children who completed the study, 83 had completed all measures a follow-up)
Not Completed | 45

BASELINE CHARACTERISTICS:
Arm/Group | ECE Center Changes Between Baseline and Follow-up
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 37
  Race: African American | 7
  Race: Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Changes in Objective Child Physical Activity
Description: Physical activity will be measured with a 7 day accelerometer at baseline and 1 year, including minutes/day MVPA in childcare center, minutes/day MVPA total. Physical activity and time spent in moderate to vigorous physical activity will be measured by a triaxial accelerometer (Actigraph GT3X+, Actigraph of Ft. Walton Beach, FL). Children will be measured on 7 full days during the baseline and follow-up periods.The Actigraph is one of the most common accelerometers used for scientific purposes, and the GT3X+ version provides extensive data on steps/day and time spent in various activity intensities. The research team will ask the parents to have the children wear the accelerometer for additional days (to a maximum of 14 days) to ensure that minimal data requirements are met.
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ECE Center Changes Between Baseline and Follow-up
Number analyzed (Participants) | 49
minutes
  Active Opportunities | 3.3 (4.1)
  Sedentary Opportunities | -0.4 (2.6)
  Sedentary Opportunities - Revised | 1.1 (4.7)
  Sedentary Environment | 0.0 (4.7)
  Portable Play Environment | 1.9 (4.0)
  Fixed Play Environment | -1.0 (4.0)

2. Secondary Outcome: Changes in Classroom Observation of Child Screen-time
Description: Classroom observation of child screen-time will be measured with the Environment and Policy Assessment and Observation (EPAO) method to quantify average minutes/day screen-time in childcare center. Screen time will be assessed using classroom observation at the childcare center (from the EPAO observation in Aim 1). Results are reflecting changes in screen-time.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | ECE Center Changes Between Baseline and Follow-up
Number analyzed (Participants) | 49
minutes/day
  Television viewing | -2.8 (8.3)
  Non-television screen-time | -18.1 (32.7)
  Total screen-time | -20.9 (39.2)

3. Secondary Outcome: Parent Reports of Child Screen Time
Description: Parent reports of child screen time to quantify minutes/day screen-time total. Parents will complete a survey adapted to provide information about the child's screen-time (separately for TV, computer, games console and smartphone) on weekdays and weekend days. For each item the parent will be asked to report the time the child spent using it for (a) a normal weekday and (b) a normal weekend day, with response options: none; 1 to 30 minutes; 31 minutes to 1 hour; 1 to 2 hours; 2 to 3 hours; 3 to 4 hours; 4 hours or more. The assessment of TV viewing using parental report has been shown to correlate moderately (r=0.60) with 10 days of TV diaries among young children.
Time Frame: 1 Year
Population: 110 parents completed the screen time survey in year 1. In Year 2 this dropped to 36. Some questions only one or two parents did not answer. All questions
Measure: Count of Participants; unit: Participants
Groups:
- Baseline; Follow-up: Parent screen report.
Arm/Group | Baseline | Follow-up
Number analyzed (Participants) | 110 | 36
Participants
  Monthly average of tv hours/day outside of school.: Less than 1 hour | 18 | 4
  Monthly average of tv hours/day outside of school.: 1 hour | 27 | 12
  Monthly average of tv hours/day outside of school.: 2 hours | 30 | 12
  Monthly average of tv hours/day outside of school.: 3 hours | 24 | 6
  Monthly average of tv hours/day outside of school.: 4 hours | 2 | 1
  Monthly average of tv hours/day outside of school.: 5 hours | 8 | 1
  Monthly average of tv hours/day outside of school.: More than 5 hours | 0 | 0
  Monthly average of tv hours/day outside of school.: None, my child does not watch TV or videos | 1 | 0
  Monthly average of computer hours/day outside of school.: Less than 1 hour | 37 | 9
  Monthly average of computer hours/day outside of school.: 1 hour | 9 | 4
  Monthly average of computer hours/day outside of school.: 2 hours | 10 | 1
  Monthly average of computer hours/day outside of school.: 3 hours | 7 | 0
  Monthly average of computer hours/day outside of school.: 4 hours | 3 | 0
  Monthly average of computer hours/day outside of school.: 5 hours | 2 | 1
  Monthly average of computer hours/day outside of school.: More than 5 hours | 0 | 0
  Monthly average of computer hours/day outside of school.: None, my child does not watch TV or videos | 42 | 21
  Monthly average of video games outside of school.: Less than 1 hour | 35 | 10
  Monthly average of video games outside of school.: 1 hour | 8 | 1
  Monthly average of video games outside of school.: 2 hours | 8 | 1
  Monthly average of video games outside of school.: 3 hours | 2 | 1
  Monthly average of video games outside of school.: 4 hours | 2 | 0
  Monthly average of video games outside of school.: 5 hours | 1 | 1
  Monthly average of video games outside of school.: More than 5 hours | 0 | 0
  Monthly average of video games outside of school.: None, my child does not watch TV or videos | 54 | 22
  Monthly average of smartphone use hours/day outside of school.: number analyzed (Participants) | 110 | 35
  Monthly average of smartphone use hours/day outside of school.: Less than 1 hour | 41 | 19
  Monthly average of smartphone use hours/day outside of school.: 1 hour | 20 | 4
  Monthly average of smartphone use hours/day outside of school.: 2 hours | 10 | 2
  Monthly average of smartphone use hours/day outside of school.: 3 hours | 5 | 1
  Monthly average of smartphone use hours/day outside of school.: 4 hours | 3 | 0
  Monthly average of smartphone use hours/day outside of school.: 5 hours | 3 | 1
  Monthly average of smartphone use hours/day outside of school.: More than 5 hours | 0 | 0
  Monthly average of smartphone use hours/day outside of school.: None, my child does not watch TV or videos | 28 | 8
  Monthly average of ipad/tablet use hours/day outside of school.: Less than 1 hour | 35 | 14
  Monthly average of ipad/tablet use hours/day outside of school.: 1 hour | 19 | 5
  Monthly average of ipad/tablet use hours/day outside of school.: 2 hours | 16 | 2
  Monthly average of ipad/tablet use hours/day outside of school.: 3 hours | 6 | 2
  Monthly average of ipad/tablet use hours/day outside of school.: 4 hours | 5 | 0
  Monthly average of ipad/tablet use hours/day outside of school.: 5 hours | 5 | 2
  Monthly average of ipad/tablet use hours/day outside of school.: More than 5 hours | 0 | 0
  Monthly average of ipad/tablet use hours/day outside of school.: None, my child does not watch TV or videos | 24 | 11

4. Secondary Outcome: Sedentary Behavior and Physical Activity
Description: Cross-sectional and longitudinal associations among sedentary behavior (by screen-time observation/self-report and accelerometry) and physical activity (by accelerometry). The mean and standard deviation for time sedentary behavior and physical activity are presented in the table below.
Time Frame: 1 year
Population: 107 participants had complete physical activity and screen-time data sets at Baseline. Researchers followed up a year later- at this follow-up time, 53 participants had complete data sets at baseline and follow-up. "Cross-sectional" arm presents the mean number of hours participants spent in light physical activity, moderate-to-vigorous physical activity, and screen time - at baseline. The "Longitudinal" arm presents means at follow-up.
Measure: Mean (Standard Deviation); unit: hours per day
Groups:
- Baseline ("Cross-sectional"); Follow-up ("Longitudinal"): Mean (SD) of Light, Moderate, Vigorous PA (hrs/day)
Arm/Group | Baseline ("Cross-sectional") | Follow-up ("Longitudinal")
Number analyzed (Participants) | 107 | 53
hours per day
  Light Physical Activity (LPA) | 4.2 (0.6) | 4.1 (0.5)
  Moderate-Vigorous Physical Activity (MVPA) | 1.7 (0.6) | 1.7 (0.5)
  Screen-time | 4.5 (3.3) | 3.8 (3.5)

5. Secondary Outcome: Fundamental Motor Skills
Description: Cross-sectional and longitudinal associations among Test of Gross Motor Development, 3rd edition (TGMD-3), and subscales (Ball Skills and Locomotor Skills). The TGMD-3 is a process-oriented assessment designed to assess gross motor performance of young children age 3-10 years. The total score for each item is established by the summation of all performance criteria scores for both trials, which are accumulated to determine the total locomotor and ball skills subtest scores and the overall TGMD-3 raw score for gross motor performance The maximum score a participant can obtain on locomotor is 46, for ball skills its 54, and overall gross motor performance is 100. The minimum score a child can receive is 0. Higher scores indicate better performance. Lower scores help identify delays and deficits in gross motor development in early childhood.
Time Frame: 1 year
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Raw Score
Groups:
- Baseline ("Cross-sectional"); Follow-up ("Longitudinal"): Mean (SD) Score of Locomotor skills, Ball skills, and overall gross motor.
Arm/Group | Baseline ("Cross-sectional") | Follow-up ("Longitudinal")
Number analyzed (Participants) | 107 | 53
Raw Score
  Locomotor Skills | 34.9 (22.8) | 35.0 (24.3)
  Ball Skills | 52.5 (24.2) | 50.9 (26.9)
  Total TGMD-3 | 41.7 (22.5) | 41.4 (23.8)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | ECE Center Changes Between Baseline and Follow-up
All-Cause Mortality (participants affected / at risk) | 0/112
Serious Adverse Events (participants affected / at risk) | 0/112
Other Adverse Events (participants affected / at risk) | 0/112

LIMITATIONS AND CAVEATS:
The timing of some assessments occurred into 2017 due to delays, there's a chance ECE centers changed their policy after the regulations were first released thus the baseline data collection was not a true baseline. However, this study did utilize handbooks for policy scoring & baseline policies were dated for the 2016-2017 school year. Another limitation is that ECE centers were aware of the day of observation, there's a potential the center made changes to present as a healthier environment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT02751814/Prot_SAP_000.pdf